CLINICAL TRIAL: NCT02547883
Title: Mortality and Economic Impact of Stopping Statins in People Aged of 75 and Over: a Pragmatic Clinical Trial
Brief Title: Statins In The Elderly
Acronym: SITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2014/41; PRME 14-0037 (Other Grant/Funding Number: French minister of Health)
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mortality
Keywords: Statins; Elderly; Mortality; Quality of life; Randomized trial; Cost effectiveness study; Primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients stopping statin (Experimental)
  Interventions: Drug: Cessation of statin
- Patients continuing statin (No Intervention)

INTERVENTIONS:
Drug: Cessation of statin — The intervention evaluated is the cessation of statin
  Arms: Patients stopping statin

SUMMARY:
In patients ≥ 75 years, there is no evidence that statins in primary prevention are associated with a decreased mortality and recent US recommendations consider statins in people only between 40 and 75 years. Moreover, statins are associated with numerous side effects impacting quality of life of those people and represent a high cost for the French healthcare system.

The aim of the present study is to evaluate cost/effectiveness ratio, in real life, of statin cessation in people ≥ 75 years treated in primary prevention.

DETAILED DESCRIPTION:
Statins in primary prevention are associated with a 1.2% decreased absolute risk of cardiovascular events in large randomized studies. Anyway, in patients ≥ 75 years, the impact of statins on mortality have not been demonstrated and large observational studies have shown an increased risk of mortality in people with low cholesterol. Moreover, statins are associated with numerous side effects, particularly in the elderly including myalgia and myositis, diabetes, cognitive disorders, fatigue and loss of energy and of physical activities, treatment interactions. At last, the cost of statins for the French national health insurance is 800 million euros per year (including around 200 million euros for people ≥ 75 years).

The benefit/risk ratio of statins is not established in primary prevention in people ≥ 75 years, leading to numerous and discordant expert advices since no specific randomized trial have been conducted in this population.

Thus, in patients ≥ 75 years treated with statins in primary prevention, the studied strategy will be to stop statin therapy. The comparison strategy will be represented by the group of patient who will continue their statin at the same dose.

Patients will be followed up every three months, according to general recommendations, during 36 months. Clinical events will be prospectively registered

ELIGIBILITY:
Inclusion Criteria:

* People aged ≥ 75 years
* Treated with any statin from at least one year, in primary prevention
* Having replied to a standardized questionnaire allowing to screen any history of cardiovascular event
* Consent form signed

Exclusion Criteria:

* Life prognosis below 6 months
* Patient with known homozygous or double heterozygous familial hypercholesterolemia
* Dementia

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Incremental Cost per QALY gained | 36 month after inclusion
  Ratio between QALYs (quality-adjusted life years) gained estimated by the EQ-5D scale and cost for the French healthcare system
Overall mortality | 36 month after inclusion

SECONDARY OUTCOMES:
Quality of life | 3, 12, 24 and 36 moth after inclusion
  Quality of life as measured by the SF12
Clinical events occurence | 3, 12, 24 and 36 moth after inclusion
  Clinical events: cardiovascular events, diabetes, cognitive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, Study Chair — USMR - CHU de Bordeaux; Jean-philippe JOSEPH, Pr, Principal Investigator — University of Bordeaux; Fabrice BONNET, Pr, Study Director — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Bonnet F, Benard A, Poulizac P, Afonso M, Maillard A, Salvo F, Berdai D, Salles N, Rousselot N, Marchi S, Hayes N, Joseph JP. Discontinuing statins or not in the elderly? Study protocol for a randomized controlled trial. Trials. 2020 Apr 19;21(1):342. doi: 10.1186/s13063-020-04259-5. PMID 32307005
- [Derived] Bonnet F, Poulizac P, Joseph JP. Safety and efficacy of statins. Lancet. 2017 Mar 18;389(10074):1097-1098. doi: 10.1016/S0140-6736(17)30712-2. No abstract available. PMID 28322812